CLINICAL TRIAL: NCT00719485
Title: A Prospective Randomized Control Trial Assessing the Effect of Two Different Educational Programs on Functional Outcome and Quality of Life Scores for Patients Having Posterior Decompressive Lumbar Spinal Surgery for Degenerative Conditions of the Lumbar Spine
Brief Title: A Study on the Use of Educational Programs Prior to Lumbar Spinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Albert Yee, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Yee_1
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2008-07

CONDITIONS: Decompression, Surgical
Keywords: lumbar decompression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Educational program
  Interventions: Other: Educational program
- 2 (No Intervention): Standard care

INTERVENTIONS:
Other: Educational program — Informing patients about their condition, treatment options, prioritization on the wait list, and post-operative care
  Arms: 1

SUMMARY:
This study evaluated the hypothesis that the implementation of an educational program that informs spine patients about their condition, treatment options, prioritization on the wait list, and post-operative care would improve functional outcome and quality of life scores following surgery

DETAILED DESCRIPTION:
Previous literature has shown that longer waits to lumbar spine surgery can have negative effects on the patients perceived function and quality of life both pre- and post-operatively. Patients report deterioration during this long wait, commonly over 6 months in Ontario. The proposed study intends to evaluate the impact of two different educational methods for patients undergoing lumbar spine surgery. This prospective randomized clinical trial will assign patients to two different educational groups: one of solely standard care, and the other of standard care with the addition of presentation of a 10 minute educational video informing spine patients about their condition, treatment options, prioritization on the wait list and post-operative care. Outcome measures will be assessed through four different questionnaires concerning specific conditions, pain, quality of life, etc., both pre-operatively and post-operatively. Providing patients with this accurate information may coincide with positive outcome measures. The more successful educational program, as found by this study, may then be provided to all spine patients. This educational program may bring about an increase in overall well-being of spine patients by having a positive impact on the quality of life both pre- and post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative condition of the lumbar spine requiring decompressive surgery

Exclusion Criteria:

* emergent spinal condition
* acute bowel/bladder dysfunction
* cervical spine condition
* inability to participate in follow up and/or functional tests or questionnaires during study timeline (due to substance abuse, etc...)
* revision surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Functional outcome scores | 2 years following surgery

SECONDARY OUTCOMES:
Quality of life scores | 2 years following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yee, MD, Principal Investigator — Sunnybrook Health Sciences Centre